CLINICAL TRIAL: NCT06275334
Title: Dinutuximab Beta at the Strasbourg University Hospitals (HUS) and the Toulouse Oncopole: Comparative Analysis of Patient Pathways, Associated Costs and Quality of Life According to Traditional Hospitalization or Hospital at Home (HAD)
Brief Title: Dinutuximab Beta at the HUS and the Toulouse Oncopole
Acronym: DNB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9133
Record Dates: First submitted 2024-02-01; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Dinutuximab Beta; DNB
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators wish to describe the cohort of pediatric patients suffering from neuroblastoma and treated with Dinutuximab and to compare the costs and quality of life between the two French centers, the University Hospital of Strasbourg (HUS) and the Oncopole of Toulouse.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 2 years to 25 years
* Male or female gender
* Subjects suffering from neuroblastoma and treated at the HUS or at the Oncopole center in Toulouse during the period from January 1, 1998 to December 31, 2023.
* Subject (and/or holders of parental authority) not opposing, after information, the reuse of the child's data for the purposes of this research and agreeing to respond to the quality of life survey.

Exclusion Criteria:

* Patient or parents of the minor having expressed their opposition to participating in the study.
* specific clinical forms of the disease,
* interfering treatments and associated diseases.

Ages: 2 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects aged 2 years to 25 years suffering from neuroblastoma and treated at the HUS or at the Oncopole center in Toulouse during the period from January 1, 1998 to December 31, 2023.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Comparison of two methods of treating a pediatric pathology in two French health establishments, the HUS and the Oncopole of Toulouse. | The period concerned is from January 1, 1998 to December 31, 2023.
  This study is retrospective and consists of comparing two methods of treating neuroblastoma in two health establishments and covers the period from January 1, 1998 to December 31, 2023.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pharmacie - Stérilisation - CHU de Strasbourg - France, Strasbourg, France